CLINICAL TRIAL: NCT03414762
Title: PICO Negative Pressure Wound Therapy in Obese Women Undergoing Elective Cesarean Delivery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-0843
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cesarean Section Complications; Cesarean Wound; Dehiscence; Cesarean Wound Disruption
Keywords: cesarean section; negative-pressure wound therapy; surgical wound dehiscence; hospital readmission; surgical site infection
MeSH Terms: conditions — Surgical Wound Dehiscence; Surgical Wound Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PICO Dressing (Experimental): PICO Negative Pressure Wound Therapy (Smith and Nephew Healthcare, Hull, United Kingdom) is a non-significant-risk, FDA Class II, medical device commercially available in the USA. The PICO unit is a single patient use, battery-powered, disposable unit that can provide continuous 80 - 125 mmHg negative pressure over a 5 to 7-day therapy period.
  Interventions: Device: PICO Negative Pressure Wound Therapy
- Standard Dressing (Active Comparator): The standard-of-care is consistent with the national standard for dressing Cesarean section incisions and includes, but not limited to, coverage of the sutured incision with sterile gauze and non-penetrable barrier (e.g., Tegaderm™). The non-penetrable barrier may be left in place for a minimum of 1 day and no longer than 2 days (± 4 hours) to promote epithelialization of the surgical incision edges. After the dressing is removed, the surgical site is left exposed to air to promote further healing.
  Interventions: Device: Standard Dressing

INTERVENTIONS:
Device: PICO Negative Pressure Wound Therapy — The PICO unit is a single patient use, battery-powered, disposable unit that can provide continuous 80 - 125 mmHg negative pressure over a 5 to 7-day therapy period.The dressing is applied to the wound and extra strips are placed over the outside edge to help hold the dressing in place. When the pump is turned on, air is pulled out of the dressing and excess fluid from the wound will start to enter the dressing.
  Other Names: PICO Dressing
  Arms: PICO Dressing
Device: Standard Dressing — The standard-of-care is consistent with the national standard for dressing Cesarean section incisions and includes, but not limited to, coverage of the sutured incision with sterile gauze and non-penetrable barrier (e.g., Tegaderm™). The non-penetrable barrier may be left in place for a minimum of 1 day and no longer than 2 days (± 4 hours) to promote epithelialization of the surgical incision edges. After the dressing is removed, the surgical site is left exposed to air to promote further healing
  Arms: Standard Dressing

SUMMARY:
A randomized controlled, parallel group, superiority, open-label, single-institution, Phase 3 interventional clinical trial to evaluate clinical outcomes in obese gravidas undergoing elective cesarean delivery whose wounds were dressed with the PICO Negative Pressure Wound Therapy (NPWT) versus the standard dressing. We hypothesize that the PICO NPWT will reduce the incidence of surgical site occurrences and interventions and postoperative readmissions in obese women. The study will compare surgical site occurrences and surgical incision intervention incidence within 42 +/- 10 days post cesarean delivery in obese women who have the current standard-of-care dressing versus the PICO NPWT.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study; willing and able to return for all scheduled and required study visits
* Female, aged 18 - 55 years
* BMI ≥ 35 kg/m2 in the 42 days prior to surgery
* In good general health as evidenced by medical history with a 24 - 41 weeks gestational age pregnancy scheduled for cesarean delivery for any routine indication (repeat procedure, breech presentation, abnormal placentation, uterine anomaly, maternal medical condition, or elective)
* Surgical skin site preparation with chlorhexidine gluconate solution (ChloraPrep©)
* Received preoperative surgical prophylaxis antibiotics as per protocol
* Surgical incision that can be covered completely by the NPWT skin system
* Pre-operatively assessed to undergo a procedure with a CDC Wound Classification of:

  a. Class I (Clean): An uninfected operative wound in which no inflammation is encountered and the respiratory, alimentary, genital, or uninfected urinary tract is not entered
* OR - b. Class II (Clean Contaminated): An operative wound in which the respiratory, alimentary, genital, or uninfected urinary tract are entered under controlled conditions and without unusual contamination
* Wound hemostasis has been achieved

Exclusion Criteria:

* Cesarean delivery before fetal viability (24 0/7 weeks gestational age)
* Unplanned Cesarean delivery
* Intrauterine fetal demise
* Known allergic reactions to components of the PICO NPWT system
* Systemic bacterial or fungal infection at the time of surgery
* Diagnosis of systemic or remote-site skin infections at time of delivery
* Treatment with another investigational drug or other intervention within 7 days prior to cesarean delivery or 42 +/- 10 days after cesarean delivery
* Delivery for suspected intrauterine infection (defined as maternal fever plus one clinical criteria)
* Critical illness or immune-compromising disease (eg acquired immunodeficiency syndrome)
* Chronic steroid use
* Pre-operatively assessed to have a CDC Wound Classification of:

Class III (Contaminated): Open, fresh, accidental wounds, and/or major breaks in sterile technique or gross spillage from the gastrointestinal tract

* OR - Class IV (Dirty-Infected): Old traumatic wounds with retained devitalized tissue and those that involve existing clinical infection or perforated viscera
* High-risk for anesthesia (American Society of Anesthesiologists [ASA] class P4 - P6)
* Intra-operative hemorrhage requiring blood transfusion, disseminated-intravascular coagulopathy (DIC) or any other medical or surgical condition during the Cesarean section deemed by the investigator to pose a prohibitively high risk for surgical re-exploration
* Unable to speak or understand English, with no interpreter available.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study is being conducted on female postpartum patient.
Enrollment: 153 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Surgical Site Occurrence | 42 days
  The incidence of postoperative Surgical Site Occurrences (SSOs) up to Day 42 (+/- 10 Days) post Cesarean Section.The incidence of postoperative surgical site occurrences (SSOs) post Cesarean delivery. SSOs include:
  * Unanticipated local inflammatory response
  * Prolonged drainage
  * Fluid collection
  * Dehiscence
  * Surgical site infection (SSI)

SECONDARY OUTCOMES:
Surgical Incision Intervention | 42 days
  Incidence rate of surgical incision intervention (SII) post Cesarean delivery.
  Interventions include:
  1. - Antimicrobials for surgical site infection
  2. - Surgical drainage of the incision
  3. - Surgical incision packing
  4. - Adjunctive negative pressure therapy
  5. - Debridement
  6. - Re-operation

CONTACTS AND LOCATIONS:
Overall Officials: Gary Goldberg, MD, Study Chair — Long Island Jewish Medical Center
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Acosta S, Bjorck M, Wanhainen A. Negative-pressure wound therapy for prevention and treatment of surgical-site infections after vascular surgery. Br J Surg. 2017 Jan;104(2):e75-e84. doi: 10.1002/bjs.10403. Epub 2016 Nov 30. PMID 27901277
- [Background] ACOG Practice Bulletin No. 120: Use of prophylactic antibiotics in labor and delivery. Obstet Gynecol. 2011 Jun;117(6):1472-1483. doi: 10.1097/AOG.0b013e3182238c31. No abstract available. PMID 21606770
- [Background] Bilgi A, Zumrut Biber Muftuler F, Akman L, Ilker Medine E, Tonbaklar Bilgi P, Kozgus Guldu O, Goksun Gokulu S, Tekin V, Cosan Terek M. In Vitro Determination of Wound Healing Potential of Axonge. Wounds. 2017 Jul;29(7):209-214. PMID 28759428
- [Background] Echebiri NC, McDoom MM, Aalto MM, Fauntleroy J, Nagappan N, Barnabei VM. Prophylactic use of negative pressure wound therapy after cesarean delivery. Obstet Gynecol. 2015 Feb;125(2):299-307. doi: 10.1097/AOG.0000000000000634. PMID 25569006
- [Background] Gillespie BM. Prophylactic Use of Negative Pressure Wound Therapy After Cesarean Delivery. Obstet Gynecol. 2015 Jul;126(1):214. doi: 10.1097/AOG.0000000000000937. No abstract available. PMID 26241279
- [Background] Grauhan O, Navasardyan A, Hofmann M, Muller P, Stein J, Hetzer R. Prevention of poststernotomy wound infections in obese patients by negative pressure wound therapy. J Thorac Cardiovasc Surg. 2013 May;145(5):1387-92. doi: 10.1016/j.jtcvs.2012.09.040. Epub 2012 Oct 27. PMID 23111014
- [Background] Leth RA, Uldbjerg N, Norgaard M, Moller JK, Thomsen RW. Obesity, diabetes, and the risk of infections diagnosed in hospital and post-discharge infections after cesarean section: a prospective cohort study. Acta Obstet Gynecol Scand. 2011 May;90(5):501-9. doi: 10.1111/j.1600-0412.2011.01090.x. Epub 2011 Mar 14. PMID 21306347
- [Background] Olsen MA, Butler AM, Willers DM, Devkota P, Gross GA, Fraser VJ. Risk factors for surgical site infection after low transverse cesarean section. Infect Control Hosp Epidemiol. 2008 Jun;29(6):477-84; discussion 485-6. doi: 10.1086/587810. PMID 18510455
- [Background] O'Leary DP, Peirce C, Anglim B, Burton M, Concannon E, Carter M, Hickey K, Coffey JC. Prophylactic Negative Pressure Dressing Use in Closed Laparotomy Wounds Following Abdominal Operations: A Randomized, Controlled, Open-label Trial: The P.I.C.O. Trial. Ann Surg. 2017 Jun;265(6):1082-1086. doi: 10.1097/SLA.0000000000002098. PMID 27926575
- [Background] Searle RJ, Myers D. A survey of caesarean section surgical site infections with PICO Single Use Negative Pressure Wound Therapy System in high-risk patients in England and Ireland. J Hosp Infect. 2017 Oct;97(2):122-124. doi: 10.1016/j.jhin.2017.02.023. Epub 2017 Aug 12. PMID 28807639
- [Background] Smid MC, Dotters-Katz SK, Grace M, Wright ST, Villers MS, Hardy-Fairbanks A, Stamilio DM. Prophylactic Negative Pressure Wound Therapy for Obese Women After Cesarean Delivery: A Systematic Review and Meta-analysis. Obstet Gynecol. 2017 Nov;130(5):969-978. doi: 10.1097/AOG.0000000000002259. PMID 29016508
- [Background] Strugala V, Martin R. Meta-Analysis of Comparative Trials Evaluating a Prophylactic Single-Use Negative Pressure Wound Therapy System for the Prevention of Surgical Site Complications. Surg Infect (Larchmt). 2017 Oct;18(7):810-819. doi: 10.1089/sur.2017.156. Epub 2017 Sep 8. PMID 28885895
- [Background] Yu L, Kronen RJ, Simon LE, Stoll CRT, Colditz GA, Tuuli MG. Prophylactic negative-pressure wound therapy after cesarean is associated with reduced risk of surgical site infection: a systematic review and meta-analysis. Am J Obstet Gynecol. 2018 Feb;218(2):200-210.e1. doi: 10.1016/j.ajog.2017.09.017. Epub 2017 Sep 23. PMID 28951263

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT03414762/Prot_000.pdf
  • Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT03414762/ICF_001.pdf